CLINICAL TRIAL: NCT04763239
Title: Prognostic Significance of Red Blood Cell Distribution Width (RDW) in Critically Ill Pediatric Patients at Sohag University Hospital
Brief Title: Prognostic Significance of Red Blood Cell
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, rezk atalla massoud, Principal Investigator, Sohag University
Other Study IDs: Soh-Med-21-02-14
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Red blood cell (RBC) distribution width (RDW), calculated by dividing the standard deviation of RBC volume by the mean corpuscular volume and multiplied by 100, is routinely reported as part of the complete blood count (CBC) using automated flow cytometry. RDW has been traditionally used as additional information in the differential diagnosis of the cause of anemia.

RDW has been recently reported as a strong prognostic factor in several diseases of various organ systems, including the cardiovascular, respiratory, renal, neurologic, and gastrointestinal systems.It also showed significant associations with ventilator-free days, postoperative outcome, intensive care unit (ICU) discharge outcome, out-of-hospital outcome, and all-cause mortality in critically ill patients. However, most studies were conducted in adult patients. Only a few studies have investigated RDW in children, especially in the critically ill pediatric population.

DETAILED DESCRIPTION:
The aim of this study is to know the prognostic significance of red blood cell distribution width ( RDW ) in critically ill pediatric patients as regard ; the duration of hospital & PICU admission ,the use of inotropic drugs and or mechanical ventilation (MV) and the outcome of the case .

ELIGIBILITY:
Inclusion Criteria:

* All critically ill pediatric patients, 1 month to 12 years age, admitted to Pediatric intermediate & Intensive Care Unit ( PICU ) in Sohag University Hospital.

Exclusion Criteria:

* - patients who received blood transfusion prior to admission in PICU
* patients with incomplete data for pediatric risk of mortality (PRISM), pediatric sequential organ failure assessment (pSOFA), pediatric logistic organ dysfunction-2 (PELOD-2), and pediatric multiple organ dysfunction syndrome (pMODS) scores were excluded.

Ages: 1 Month to 12 Years | Sex: All
Age Groups: Child
Study Population: All patients included in this study will be subjected to the following (as detailed in the attached patient's data sheet).
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
duration of hospital admission | 6 months
  in days

CONTACTS AND LOCATIONS:
Overall Officials: shimaa mahmoud, Professor, Study Director — Sohag University
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weiss G, Goodnough LT. Anemia of chronic disease. N Engl J Med. 2005 Mar 10;352(10):1011-23. doi: 10.1056/NEJMra041809. No abstract available. PMID 15758012
- [Background] Jo YH, Kim K, Lee JH, Kang C, Kim T, Park HM, Kang KW, Kim J, Rhee JE. Red cell distribution width is a prognostic factor in severe sepsis and septic shock. Am J Emerg Med. 2013 Mar;31(3):545-8. doi: 10.1016/j.ajem.2012.10.017. Epub 2013 Feb 4. PMID 23380094